CLINICAL TRIAL: NCT05266742
Title: Investigation of the Effect of Web-based Education on Self-Care Management and Family Support in Women With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, Ceren Dilek MUMCU, Principal Investigator, PhD student, RN, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AnkaraYBU132435
Record Dates: First submitted 2022-01-20; First posted 2022-03-04 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Diabetes Type 2
Keywords: Diabetes Mellitus; nurse; self care; web based education; family
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- END (Experimental): Use of web based education
  Interventions: Other: web based education
- END free (No Intervention): patient witout of web based education

INTERVENTIONS:
Other: web based education — An educative website was created for our study. The content of the website was accessible from "www.diyabet.mumcu.net" and the content of the website was brought together by scanning the literature. The content text was quoted from publicly available information and guides as ADA and IDF.
  Arms: END

SUMMARY:
This is a quasi-experimental study that was carried out to examine the effect of the web-based education given to female individuals using insulin with Type 2 diabetes on self-care management and family support.

Methods A randomized controlled trial using a sample (N=66) of women with type 2 diabetes who admitted to the hospital's outpatient clinic in 2020. The intervention group received web-based education for six months. Socio-demographic data, metabolic values, "Diabetes Self-Care Scale" and "Family Support and Conflict Scale in Type 2 Diabetes" were used.

DETAILED DESCRIPTION:
Methods This quasi-experimental study was conducted in Ankara, Turkey, 2020. Sixty six patients were selected using convenient sampling and divided equally into two control and intervention groups based on random allocation. Web-based education was provided to the intervention group for six months. Data were collected before, at the third month of the intervention, and at the end of the intervention using "Patient Identification Form", "Metabolic Control Variables Form", "Diabetes Self-Care Scale" and "Family Support and Conflict Scale in Type 2 Diabetes" forms. All the patients were female individuals diagnosed with Type 2 diabetes at least a year ago, using insulin between the ages of 18 to 65 years old, who applied to the internal medicine and endocrine outpatient clinic of a training and research hospital in Ankara. Patients had no communication barriers, and they were able to use computers and smartphones and volunteer for this study. No consultancy training was given to the control group by the researcher. They only received routine education in the hospital.

Data Collection Tools Data is collected using "Patient Identification Form", "Metabolic Control Variables Form", "Diabetes Self-Care Scale" and "Family Support and Conflict Scale in Type 2 Diabetes" forms.

Patient Identification Form Patient Identification Form was created for this study by scanning the literature. In this form, there were 12 questions in total. The questions included the first letters of the name and surname for coding purposes. There were questions about the age, marital status, employment status, educational status, smoking, alcohol and snacking habits, regular insulin use, blood glucose measurement, physical activity, dietary compliance, and previous educations about diabetes.

Metabolic Control Variables Form Metabolic Control Variables Form was created for this study by scanning the literature. It had questions regarding the disease of the individuals. The questions were about fasting blood glucose, HbA1c, LDL, HDL, total cholesterol, triglycerides, weight, height, and body mass index.

Diabetes Self-Care Scale Diabetes Self-Care Scale is a survey. Diabetes Self-Care Scale was developed by Lee and Fisher in 2005. It aims to evaluate the self-care activities of patients with type 2 diabetes. This scale was adapted and translated to Turkish by Karakurt and Kaşıkçı in 2008. The options of the scale were changed to "Never (1)" "Sometimes (2)" "Frequently (3)" and "Always (4)". It has been stated that patients who score points more than 66% of the scale total points are assumed at a level to meet their self-care. Based on the 4-point Likert type, the maximum score of the scale was 140 points. As the score increases, the self-care activities of the patients increase positively. Diabetes Self-Care Scale contains 35 items. The scale does not have sub-dimensions and inverse expressions. These items aim to get information about eating on time, exercising, measuring and recording blood sugar, using oral antidiabetics and insulin as recommended, visiting a doctor for checking blood sugar, foot care, personal hygiene practices, diabetes, and its complications. While the Cronbach Alpha value of the scale developed by Lee and Fisher was determined to be 0.80, the total Cronbach Alpha coefficient of the scale in Karakurt's research was determined as 0.81.

Family Support and Conflict Scale in Type 2 Diabetes The Family Support and Conflict Scale in Type 2 Diabetes is a survey. The Family Support and Conflict Scale in Type 2 Diabetes was prepared by Charlotte Paddison in Japan in 2010 for individuals with type 2 diabetes. It consists of informative questions about the support status of the family and conflicts with the family. The scale was adapted to Turkish by Sofulu and Avdal in 2015 and the Cronbach Alpha coefficient of the scale is 0.740. DFSC has two sub-dimensions being 'Family Support' and 'Family Conflict'. The highest score obtained from the sub-dimensions was 50 and the lowest score was 10. As the subscale scores increase, the level of support increases. As the family conflict sub-dimension score decreases, the family conflict increase. The answers in the scale are 5-point Likert type and are classified as strongly agree, agree, undecided, disagree, strongly disagree. The scale contains 10 items in total. The items aim to get information to measure the family's attitude towards the diet, exercise, medications, and mental state of the diabetic.

Website An educative website was created for our study. The content of the website was accessible from "www.diyabet.mumcu.net" and the content of the website was brought together by scanning the literature. The content text was quoted from publicly available information and guides as ADA and IDF. The pictures on the website were obtained from license-free sources. The website also included a training video that was prepared by the researcher. The website was developed by using Microsoft Asp.NET MVC technology and it was designed responsively for ease of use. The website could be accessed from computers, tablets, and smartphones. Expert opinions were obtained using the DISCERN Measurement Tool to evaluate the reliability and quality of the training material. A username and a password were provided separately for each of the 33 individuals in the intervention group. In addition to the user content, the website had a separate management panel that was only used by the researcher. Using this admin panel, the researcher could see the pages that the participants in the intervention group accessed on the website, and the page visit times were available in logs. The content of the website is divided into training modules. These modules were published to the users sequentially during six months period by allowing access to a new module a month. A reminder message was sent twice a week to the user regarding the subject of the training module.

Application of Data Collection Tools Patient identification form, metabolic control variables form, Diabetes Self-Care Scale and Family Support and Conflict Scale in Type 2 Diabetes were administered face-to-face with interviews to the individuals included in the study when they came to their outpatient clinic appointments. In the third month of the study, the laboratory results of the hospital system were obtained and the form of metabolic control variables was recorded. It has been obtained from the routine laboratory results that were checked every three months upon the doctor's request. No blood was taken from individuals by the researcher. Web-based education was provided to the intervention group for six months. The metabolic control variables form, Diabetes Self-Care Scale and Family Support and Conflict Scale in Type 2 Diabetes were administered by the researcher using face-to-face interviews, e-mails, and mobile phone calls to the intervention and control groups based on their request at the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with Type 2 diabetes at least a year ago
* using insulin
* able to use computers and smartphones

Exclusion Criteria:

* Not having been diagnosed with diabetes

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2019-12-15 (Actual); Primary Completion 2020-05-15 (Actual); Study Completion 2020-08-15 (Actual)

PRIMARY OUTCOMES:
Diabetes Self-Care Scale | a day before the education
  Diabetes Self-Care Scale Diabetes Self-Care Scale is a survey. It has been stated that patients who score points more than 66% of the scale total points are assumed at a level to meet their self-care. Based on the 4-point Likert type, the maximum score of the scale was 140 points. As the score increases, the self-care activities of the patients increase positively. It contains 35 items. These items aim to get information about eating on time, exercising, measuring and recording blood sugar, using oral antidiabetics and insulin as recommended, visiting a doctor for checking blood sugar, foot care, personal hygiene practices, diabetes, and its complications.
Family Support and Conflict Scale in Type 2 Diabetes | a day before the education
  The Family Support and Conflict Scale in Type 2 Diabetes is a survey. DFSC has two sub-dimensions being 'Family Support' and 'Family Conflict'. The highest score obtained from the sub-dimensions was 50 and the lowest score was 10. As the subscale scores increase, the level of support increases. As the family conflict sub-dimension score decreases, the family conflict increase. The answers in the scale are 5-point Likert type and are classified as strongly agree, agree, undecided, disagree, strongly disagree. The scale contains 10 items in total. The items aim to get information to measure the family's attitude towards the diet, exercise, medications, and mental state of the diabetic.
Metabolic Control Variables Form | a day before the education
  Metabolic Control Variables Form is created for this study by scanning the literature. It has questions regarding the disease of the individuals. The questions are about fasting blood glucose, HbA1c, LDL, HDL, total cholesterol, triglycerides, weight, height, and body mass index.
Patient Identification Form | a day before the education
  Patient Identification Form is created for this study by scanning the literature. In this form, there are 12 questions in total. The questions included the first letters of the name and surname for coding purposes. There are questions about the age, marital status, employment status, educational status, smoking, alcohol and snacking habits, regular insulin use, blood glucose measurement, physical activity, dietary compliance, and previous educations about diabetes.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No